CLINICAL TRIAL: NCT04063007
Title: The Potential Impact of the Ketogenic Diet on Epigenetics and Gut Microbiota in Children With Epilepsy
Brief Title: Epigenetics and Gut Microbiota in Children With Epilepsy
Acronym: EpiMICRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian University of Life Sciences (Other); University of Oslo (Other); Lund University (Other)
Responsible Party: Principal Investigator, Kaja Kristine Selmer, Senior Scientist, MD, PhD, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016/2016/REK sør-øst
Record Dates: First submitted 2018-11-11; First posted 2019-08-20 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: This is a prospective, non-randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketogenic diet (Other): The patients follow the ordinary treatment protocol for initiation and follow-up of the ketogenic diet
  Interventions: Other: Ketogenic diet

INTERVENTIONS:
Other: Ketogenic diet — The patients follow the ordinary treatment protocol for ketogenic diet

SUMMARY:
The ketogenic diet is a high-fat, low-carbohydrate diet used in the treatment of epilepsy. The diet can be an efficient treatment option in children with drug resistant epilepsy, with more than 50 % seizure reduction in about 40- 70 % of the patients. However, there is still a lack of knowledge regarding the mechanisms of action, how will respond to the treatment and potential adverse effects.

DETAILED DESCRIPTION:
The ketogenic diet is a high-fat, moderate protein, low-carbohydrate diet. It is an internationally established treatment option in children with drug resistant epilepsy. About 40 -70 % of children with drug resistant epilepsy treated with the ketogenic diet achieve > 50 % seizure reduction. However, even though the ketogenic diet has been used in the treatment of epilepsy for almost a Century, little is known about how the dietary treatment reduces seizures and which patients that will respond well. In addition, there is limited knowledge about potential adverse effects of the treatment. This is a prospective study following the patients from 4 weeks before initiating the ketogenic diet and during the treatment. The influence of the dietary treatment on the gut microbiota, epigenetics, quality of life, and adverse effects will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Drug resistant epilepsy
* Age 2- 17 years
* Two or more countable seizures/week
* Willing to try treatment with the ketogenic diet for at least 12 weeks

Exclusion Criteria:

* Glucose transporter protein 1 deficiency, pyruvate dehydrogenase deficiency, or pyruvate carboxylase deficiency
* Known or suspected disease in wich the diet is contraindicated
* Epilepsy surgery the last 6 months before diet initiation
* Steroid medications the last 2 months before diet initiation
* Breastfeeding
* Psychogenic non-epileptic seizures
* Eating disorder
* Pregnancy or planed pregnancy
* Feeding disabilities not compatible with dietary treatment
* Inability to follow study scheme
* Previous treatment with high-fat, low- carbohydrate diet
* Medical need to start dietary treatment immediately

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2017-08-15 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Characterization of the gut microbiota | From baseline to 12 weeks of dietary treatment.
  Changes in the gut microbiota composition in fecal samples from baseline to 12 weeks of dietary treatment will be measured by 16S rRNA analysis.
Characterization of DNA methylation | From baseline to 12 weeks of dietary treatment.
  Changes in the DNA methylation in white blood cells from baseline to 12 weeks of dietary treatment will be analyzed using the Infinium Methylation EPIC Kit.

SECONDARY OUTCOMES:
Changes in parental quality of life and parental perceptions of their child's quality of life | 12 weeks of dietary treatment.
  The impact of the dietary treatment on quality of life will be examined by using a questionaire before and after 12 weeks of dietary treatment. The quality of life score is a parental measure of the impact for the family, based on their hopes and expectations of the effects of the ketogenic diet.The quality of life is rate on a scale from 0 to 10 (0 = quality of life is poor, 10 = quality of life is very good)
Adverse effects | 12 weeks of dietary treatment.
  To identify potential adverse effects induced by the dietary treatment measured by a structured interview.

CONTACTS AND LOCATIONS:
Overall Officials: Kaja K Selmer, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided